CLINICAL TRIAL: NCT04646148
Title: Optimization and Multi-Site Feasibility of Yoga for Chronic Pain in People in Treatment for Opioid Use Disorder - Phase I
Brief Title: Optimization and Multi-Site Feasibility of Yoga for Chronic Pain in People in YOGAMAT-II - Phase I
Acronym: YOGAMAT-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: 202002-002-1; U01AT010863 (NIH)
Record Dates: First submitted 2020-11-12; First posted 2020-11-27 (Actual); Results first posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-08

CONDITIONS: Opioid Use; Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- No Video/No One-on-One/No Text/No Incentive (Active Comparator): This group does not receive Personal Practice Videos, or One-on-One individual sessions with a Yoga Instructor, or prompting Text messages, or financial Incentives to attend yoga classes
  Interventions: Behavioral: Yoga classes
- No Video/No One-on-One/No Text/Yes Incentive (Active Comparator): This group does not receive Personal Practice Videos, or One-on-One individual sessions with a Yoga Instructor, or prompting Text messages, but DOES receive financial Incentives to attend yoga classes
  Interventions: Behavioral: Yoga classes
- No Video/No One-on-One/Yes Text/No Incentive (Active Comparator): This group does not receive Personal Practice Videos, or One-on-One individual sessions with a Yoga Instructor, or financial Incentives to attend yoga classes, but DOES recieve prompting Text messages,
  Interventions: Behavioral: Yoga classes
- No Video/No One-on-One/Yes Text/Yes Incentive (Active Comparator): This group does not receive Personal Practice Videos, or One-on-One individual sessions with a Yoga Instructor, but DOES receive prompting Text messages, and financial Incentives to attend yoga classes
  Interventions: Behavioral: Yoga classes
- No Video/Yes One-on-One/No Text/No Incentive (Active Comparator): This group does not receive Personal Practice Videos, or prompting Text messages, or financial Incentives to attend yoga classes, but DOES receive One-on-One individual sessions with a Yoga Instructor
  Interventions: Behavioral: Yoga classes
- No Video/Yes One-on-One/No Text/Yes Incentive (Active Comparator): This group does not receive Personal Practice Videos, or prompting Text messages, but DOES receive financial Incentives to attend yoga classes and One-on-One individual sessions with a Yoga Instructor
  Interventions: Behavioral: Yoga classes
- No Video/Yes One-on-One/Yes Text/No Incentive (Active Comparator): This group does not receive Personal Practice Videos, or financial Incentives to attend yoga classes, but DOES receive prompting Text messages and One-on-One individual sessions with a Yoga Instructor
  Interventions: Behavioral: Yoga classes
- No Video/Yes One-on-One/Yes Text/Yes Incentive (Active Comparator): This group does not receive Personal Practice Videos, but DOES receive financial Incentives to attend yoga classes, prompting Text messages and One-on-One individual sessions with a Yoga Instructor
  Interventions: Behavioral: Yoga classes
- Yes Video/No One-on-One/No Text/No Incentive (Active Comparator): This group does not receive financial Incentives to attend yoga classes, prompting Text messages or One-on-One individual sessions with a Yoga Instructor, but DOES receive Personal Practice Videos
  Interventions: Behavioral: Yoga classes
- Yes Video/No One-on-One/No Text/Yes Incentive (Active Comparator): This group does not receive prompting Text messages or One-on-One individual sessions with a Yoga Instructor, but DOES receive financial Incentives to attend yoga classes and Personal Practice Videos
  Interventions: Behavioral: Yoga classes
- Yes Video/No One-on-One/Yes Text/No Incentive (Active Comparator): This group does not receive financial Incentives to attend yoga classes, or One-on-One individual sessions with a Yoga Instructor, but DOES receive Personal Practice Videos and prompting Text messages
  Interventions: Behavioral: Yoga classes
- Yes Video/No One-on-One/Yes Text/Yes Incentive (Active Comparator): This group does not receive One-on-One individual sessions with a Yoga Instructor, but DOES receive Personal Practice Videos, prompting Text messages and financial Incentives to attend yoga classes
  Interventions: Behavioral: Yoga classes
- Yes Video/Yes One-on-One/No Text/No Incentive (Active Comparator): This group does not receive prompting Text messages or financial Incentives to attend yoga classes, but DOES receive One-on-One individual sessions with a Yoga Instructor and Personal Practice Videos
  Interventions: Behavioral: Yoga classes
- Yes Video/Yes One-on-One/No Text/Yes Incentive (Active Comparator): This group does not receive prompting Text messages but DOES receive financial Incentives to attend yoga classes, One-on-One individual sessions with a Yoga Instructor and Personal Practice Videos
  Interventions: Behavioral: Yoga classes
- Yes Video/Yes One-on-One/Yes Text/No Incentive (Active Comparator): This group does not receive financial Incentives to attend yoga classes, but DOES receive prompting Text messages, One-on-One individual sessions with a Yoga Instructor and Personal Practice Videos
  Interventions: Behavioral: Yoga classes
- Yes Video/Yes One-on-One/Yes Text/Yes Incentive (Active Comparator): This group receives Personal Practice Videos, One-on-One individual sessions with a Yoga Instructor, prompting Text messages, and financial Incentives to attend yoga classes
  Interventions: Behavioral: Yoga classes

INTERVENTIONS:
Behavioral: Yoga classes — All participants are invited to attend weekly yoga classes.

SUMMARY:
Phase 1 - MOST Preparation Phase:

1. To conduct a pilot trial at two opioid use disorder clinic sites, enrolling n=10 at both sites, for a total n=20.
2. Establish clinical trial procedures and document feasibility at both sites prior to conducting a fully powered optimization trial.
3. Demonstrate our ability to a) recruit participants; b) train yoga teachers to fidelity; c) randomize participants to intervention components and correctly administer components; d) run classes; and e) collect follow-up assessments.

DETAILED DESCRIPTION:
In Phase 1, we will enroll 10 participants at each recruitment site (n=20). The purpose of Phase 1 (MOST Preparation Phase) is to allow us to establish and refine procedures at these new sites and document aspects of feasibility, including our ability to a) recruit participants; b) train yoga teachers to fidelity; c) randomize participants to intervention components and correctly administer these components; d) run classes; and e) collect follow-up assessments. Enrollment period for this phase will last approximately 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in methadone maintenance (MMT) or buprenorphine/naloxone (BUP) treatment for > 3 months
* Plan to continue treatment for next 6 months
* Chronic pain, defined as pain for at least half the days over the previous three months, a mean score of 4 or higher on the Brief Pain Interference Scale (BPI; with reference to chronic pain), and pain severity of 4 or higher on a Visual Analog Scale (0-10) indicating "worst pain in the last week." Pain severity score will also refer to the areas of their body in which they have chronic pain.
* Aged > 18
* Proficiency in English sufficient to engage in informed consent in English, understand classes taught in English, and read short sentences
* Available at least one of the times study classes are offered.

Exclusion Criteria:

* Currently taking yoga classes or practicing yoga at home once per week or more often.
* Medical conditions that would make participation in yoga unsafe or not possible, including active malignancy treatment, fracture, recent joint surgery, use of assistive ambulatory devices other than a cane. . (In cases where this is unclear, site PI will make final determination based on available evidence.)
* Severe or progressive neurologic deficits. (In cases where this is unclear, site PI will make final determination based on available evidence.)
* Other severe disabling chronic medical and/or psychiatric comorbidities deemed by the site PI on a case-by-case basis to prevent safe or adequate participation in the study (e.g., cognitive impairment that prevents a participant from understanding assessments; history of disruptive behavior in medical settings; severe disabling heart failure or lung disease)
* Surgery requiring overnight hospitalization planned in the next 3 months
* Pregnancy
* Plan to move out of the area within 6 months.
* Homeless, defined as any time in the past month sleeping in a shelter or on the street.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Boston Medical Center, Boston, Massachusetts
  - CODAC Behavioral Healthcare, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Video/No One-on-One/No Text/No Incentive | No Video/No One-on-One/No Text/Yes Incentive | No Video/No One-on-One/Yes Text/No Incentive | No Video/No One-on-One/Yes Text/Yes Incentive | No Video/Yes One-on-One/No Text/No Incentive | No Video/Yes One-on-One/No Text/Yes Incentive | No Video/Yes One-on-One/Yes Text/No Incentive | No Video/Yes One-on-One/Yes Text/Yes Incentive | Yes Video/No One-on-One/No Text/No Incentive | Yes Video/No One-on-One/No Text/Yes Incentive | Yes Video/No One-on-One/Yes Text/No Incentive | Yes Video/No One-on-One/Yes Text/Yes Incentive | Yes Video/Yes One-on-One/No Text/No Incentive | Yes Video/Yes One-on-One/No Text/Yes Incentive | Yes Video/Yes One-on-One/Yes Text/No Incentive | Yes Video/Yes One-on-One/Yes Text/Yes Incentive
Started | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 2 | 1 | 2 | 1 | 2 | 1 | 1 | 2 | 2
Completed | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 2 | 1 | 1 | 2 | 0
Not Completed | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: This was a pilot study. We planned ahead of time that some arms would not be populated.
Groups:
- Total: Total of all reporting groups
Arm/Group | No Video/No One-on-One/No Text/No Incentive | No Video/No One-on-One/No Text/Yes Incentive | No Video/No One-on-One/Yes Text/No Incentive | No Video/No One-on-One/Yes Text/Yes Incentive | No Video/Yes One-on-One/No Text/No Incentive | No Video/Yes One-on-One/No Text/Yes Incentive | No Video/Yes One-on-One/Yes Text/No Incentive | No Video/Yes One-on-One/Yes Text/Yes Incentive | Yes Video/No One-on-One/No Text/No Incentive | Yes Video/No One-on-One/No Text/Yes Incentive | Yes Video/No One-on-One/Yes Text/No Incentive | Yes Video/No One-on-One/Yes Text/Yes Incentive | Yes Video/Yes One-on-One/No Text/No Incentive | Yes Video/Yes One-on-One/No Text/Yes Incentive | Yes Video/Yes One-on-One/Yes Text/No Incentive | Yes Video/Yes One-on-One/Yes Text/Yes Incentive | Total
Number analyzed (Participants) | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 2 | 1 | 2 | 1 | 2 | 1 | 1 | 2 | 2 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 30 (0) |  | 38 (0) | 32 (0) | 48.5 (12.5) | 46 (0) | 52.5 (18.5) | 59 (0) | 54.5 (1.5) | 50 (0) | 51 (9) | 35 (0) | 59 (0) | 55 (10) | 49 (1) | 48.5 (11.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 |  | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 12
  Male |  | 0 |  | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 |  | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Not Hispanic or Latino |  | 1 |  | 1 | 1 | 1 | 0 | 2 | 1 | 2 | 1 | 2 | 1 | 1 | 2 | 2 | 18
  Unknown or Not Reported |  | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian |  | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American |  | 0 |  | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 4
  White |  | 1 |  | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 10
  More than one race |  | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3
  Unknown or Not Reported |  | 0 |  | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States |  | 1 |  | 1 | 1 | 2 | 1 | 2 | 1 | 2 | 1 | 2 | 1 | 1 | 2 | 2 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Recruited
Description: As this is a pilot study, a key outcome is number of participants recruited
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Groups:
- Entire Study: Because this outcome was a feasibility/ acceptability outcome, it is reported across the entire study.
Arm/Group | Entire Study
Number analyzed (Participants) | 20
Participants | 20

2. Primary Outcome: Number of Yoga Teachers Trained to > 80% Fidelity to the Manual
Description: As this is a pilot study, an outcome is to assess whether we can train teachers to an acceptable level of fidelity
Time Frame: 7 months
Population: 5 yoga teachers trained and taught classes
Measure: Count of Participants; unit: Participants
Arm/Group | Entire Study
Number analyzed (Participants) | 5
Participants | 4

3. Primary Outcome: Percent of Weeks Where Data on Amount of Yoga Personal Practice Were Collected
Description: As this is a pilot study, an outcome is percentage of weeks where data on amount of yoga personal practice were collected. The total number of weeks possible = 12. These data are most important as they will be used to derive the primary outcome in the next phase of this research (total amount of yoga practice.)
Time Frame: 3 months
Population: By design, no one was assigned to group 1 or 3.
Measure: Mean (Standard Deviation); unit: percentage of weeks
Arm/Group | No Video/No One-on-One/No Text/No Incentive | No Video/No One-on-One/No Text/Yes Incentive | No Video/No One-on-One/Yes Text/No Incentive | No Video/No One-on-One/Yes Text/Yes Incentive | No Video/Yes One-on-One/No Text/No Incentive | No Video/Yes One-on-One/No Text/Yes Incentive | No Video/Yes One-on-One/Yes Text/No Incentive | No Video/Yes One-on-One/Yes Text/Yes Incentive | Yes Video/No One-on-One/No Text/No Incentive | Yes Video/No One-on-One/No Text/Yes Incentive | Yes Video/No One-on-One/Yes Text/No Incentive | Yes Video/No One-on-One/Yes Text/Yes Incentive | Yes Video/Yes One-on-One/No Text/No Incentive | Yes Video/Yes One-on-One/No Text/Yes Incentive | Yes Video/Yes One-on-One/Yes Text/No Incentive | Yes Video/Yes One-on-One/Yes Text/Yes Incentive
Number analyzed (Participants) | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 2 | 1 | 2 | 1 | 2 | 1 | 1 | 2 | 2
percentage of weeks |  | 100 (0) |  | 100 (0) | 8.3 (0) | 62.5 (53.03) | 100 (0) | 58.3 (58.92) | 100 (0) | 100 (0) | 100 (0) | 100 (0) | 100 (0) | 100 (0) | 100 (0) | 12.5 (17.68)

ADVERSE EVENTS:
Time Frame: 3 months -- this is the length of time that any one participant was enrolled in the study.
Description: In some arms, # of participants at risk = 0 because 0 people were assigned to that arm in this pilot study.
Arm/Group | No Video/No One-on-One/No Text/No Incentive | No Video/No One-on-One/No Text/Yes Incentive | No Video/No One-on-One/Yes Text/No Incentive | No Video/No One-on-One/Yes Text/Yes Incentive | No Video/Yes One-on-One/No Text/No Incentive | No Video/Yes One-on-One/No Text/Yes Incentive | No Video/Yes One-on-One/Yes Text/No Incentive | No Video/Yes One-on-One/Yes Text/Yes Incentive | Yes Video/No One-on-One/No Text/No Incentive | Yes Video/No One-on-One/No Text/Yes Incentive | Yes Video/No One-on-One/Yes Text/No Incentive | Yes Video/No One-on-One/Yes Text/Yes Incentive | Yes Video/Yes One-on-One/No Text/No Incentive | Yes Video/Yes One-on-One/No Text/Yes Incentive | Yes Video/Yes One-on-One/Yes Text/No Incentive | Yes Video/Yes One-on-One/Yes Text/Yes Incentive
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1 | 0/0 | 0/1 | 0/1 | 0/2 | 0/1 | 0/2 | 0/1 | 0/2 | 0/1 | 0/2 | 0/1 | 0/1 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/0 | 0/1 | 0/1 | 0/2 | 0/1 | 0/2 | 0/1 | 0/2 | 0/1 | 0/2 | 0/1 | 0/1 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/0 | 1/1 | 0/1 | 0/2 | 0/1 | 1/2 | 0/1 | 1/2 | 0/1 | 1/2 | 1/1 | 1/1 | 2/2 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | No Video/No One-on-One/No Text/No Incentive (N=0) | No Video/No One-on-One/No Text/Yes Incentive (N=1) | No Video/No One-on-One/Yes Text/No Incentive (N=0) | No Video/No One-on-One/Yes Text/Yes Incentive (N=1) | No Video/Yes One-on-One/No Text/No Incentive (N=1) | No Video/Yes One-on-One/No Text/Yes Incentive (N=2) | No Video/Yes One-on-One/Yes Text/No Incentive (N=1) | No Video/Yes One-on-One/Yes Text/Yes Incentive (N=2) | Yes Video/No One-on-One/No Text/No Incentive (N=1) | Yes Video/No One-on-One/No Text/Yes Incentive (N=2) | Yes Video/No One-on-One/Yes Text/No Incentive (N=1) | Yes Video/No One-on-One/Yes Text/Yes Incentive (N=2) | Yes Video/Yes One-on-One/No Text/No Incentive (N=1) | Yes Video/Yes One-on-One/No Text/Yes Incentive (N=1) | Yes Video/Yes One-on-One/Yes Text/No Incentive (N=2) | Yes Video/Yes One-on-One/Yes Text/Yes Incentive (N=2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Edema in limbs (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

LIMITATIONS AND CAVEATS:
This was a pilot study that was designed to assess feasibility of the proposed design prior to starting a larger trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT04646148/Prot_SAP_000.pdf